CLINICAL TRIAL: NCT03305289
Title: Brain Activity Assessment by Functional MRI Before, After Radiofrequency of Gasserian Ganglia in Patient With Trigeminal Neuralgia
Brief Title: FMRI Assessment After Radiofrequency in Trigeminal Neuralgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed elsayed, assisstant lecture, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RF in trigeminal neuralgia
Record Dates: First submitted 2017-09-22; First posted 2017-10-09 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Trigeminal Neuralgia; Pain, Neuropathic
MeSH Terms: conditions — Trigeminal Neuralgia; Neuralgia | interventions — Pulsed Radiofrequency Treatment; Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulsed radiofrequency (Active Comparator): sensory stimulation will be carried out at 50 Hz. The definitive position of the electrode will be verified by inducing paresthesia with sensory stimulation between 0.1-0.3 V in the affected painful area, then pulsed radiofrequency will be applied for 10 patients for 10 mins
  Interventions: Procedure: pulsed Radiofrequency
- thermal Radiofrequency (Active Comparator): sensory stimulation will be carried out at 50 Hz. The definitive position of the electrode will be verified by inducing paresthesia with sensory stimulation between 0.1-0.3 V in the affected painful area, then Thermal lesion will be applied for 10 patients for 2 cycles of 90 seconds
  Interventions: Procedure: thermal Radiofrequency

INTERVENTIONS:
Procedure: pulsed Radiofrequency — sensory stimulation will be carried out at 50 Hz. The definitive position of the electrode will be verified by inducing paresthesia with sensory stimulation between 0.1-0.3 V in the affected painful area, then pulsed radiofrequency will be applied for 10 patients for 10 mins
  Arms: pulsed radiofrequency
Procedure: thermal Radiofrequency — sensory stimulation will be carried out at 50 Hz. The definitive position of the electrode will be verified by inducing paresthesia with sensory stimulation between 0.1-0.3 V in the affected painful area, then Thermal lesion will be applied for 10 patients for 2 cycles of 90 seconds
  Arms: thermal Radiofrequency

SUMMARY:
To investigate the brain activations related to TN, using fMRI, and to evaluate changes in these activations following the application of pulsed and thermal Radiofrequency lesioning to the gasserien ganglion.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 65 years
* Primary trigeminal neuralgia
* Maxillary and/or mandibular affection only
* Failure of medical treatment

Exclusion Criteria:

* 2ry trigeminal neuralgia
* Recurrent trigeminal neuralgia
* Ophthalmic branch affection
* Contraindication for intervention (sepsis, coagulopathy, infection at entery point, local anesthetic allergy,…)
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
pain alleviation | 1 month
  pain assessment by functional MRI

IPD SHARING:
Plan to Share IPD: Undecided